CLINICAL TRIAL: NCT02652793
Title: Simplification From Tenofovir Plus Lamivudine or Emtricitabine Plus Ritonavir-Boosted-Protease Inhibitor to Ritonavir-Boosted-Atazanavir Plus Lamivudine in Virologically-Suppressed-HIVInfected Adults With Osteopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Judit Pich (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Sponsor-Investigator, Judit Pich, Clinical Research Manager, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Osteosimply014; 2014-002720-27 (EudraCT Number)
Record Dates: First submitted 2015-12-31; First posted 2016-01-12 (Estimated); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): All participants will switch their current antiretroviral regimen to a boosted atazanavir and lamivudine once daily.
  Interventions: Drug: Boosted atazanavir; Drug: Lamivudine

INTERVENTIONS:
Drug: Boosted atazanavir — Atanazir 300 mg once dailly boosted with 100 mg of ritonavir once dailly
Drug: Lamivudine — Lamivudine 300 mg once dailly

SUMMARY:
A 48-week, open label, non comparative prospective trial in stable chronic human immunodeficiency virus-infected patients having achieved complete virological suppression for more than 24 weeks (human immunodeficiency virus-1 RNA <50 c/ml) switching from an antiretroviral regimen containing tenofovir and lamivudine or emtricitabine and boosted protease inhibitor to boosted atazanavir and lamivudine Study visits will take place at screening, baseline, weeks 4, 12, 24, and 48.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus-1-infected subjects with age ≥18 years old
* Hip or spine T-scores between < -1.0 and >-2.5 by dual-energy X-ray absorptiometry (in the previous 24 weeks)
* Stable antiretroviral treatment based on tenofovir and lamivudine or emtricitabine and boosted protease inhibitor for at least 24 weeks.
* Having plasma human immunodeficiency virus-1 RNA <50 copies/mL for at least the previous 24 weeks, including at least two samples.

Exclusion Criteria:

* Pregnancy, breast-feeding status or plans for pregnancy in the short term
* Primary genotypic resistance mutations and/or previous virological failures to atazanavir or lamivudine/emtricitabine
* Chronic hepatitis B infection
* Patients with indication for therapy for the prevention of bone fractures
* 25-OH vitamin D deficiency (< 10ng/mL)
* Hypogonadism (low total testosterone according to local reference range)
* Hypothyroidism (low T4 and increased thyroid stimulating hormone levels according to local reference ranges)
* Hyperparathyroidism (increased parathyroid hormone level with hypercalcaemia according to local reference ranges)
* Having received oral corticosteroids or inhaled fluticasone (daily doses higher than 5 mg/d prednisone equivalent for 3 months or more)
* Using anti-resorptive therapy (Calcium and vitamin D supplements are encouraged but not mandated)
* Body mass index lower than 19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic i Provincial de Barcelona, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center (Infectious Diseases Department, Hospital Clínic, University of Barcelona) between November 2015 and November 2017. Recruitment targeted virologically suppressed HIV-infected adults with osteopenia receiving tenofovir-based ART.
Pre-assignment Details: Of the 60 individuals screened, 29 were excluded prior to assignment due to normal bone mineral density, prior virological failure, hypogonadism, or contraindicated medications. A total of 31 participants were enrolled and switched to the study regimen.
Groups:
- RTV-Boosted-ATV + 3TC: Participants switched from a stable antiretroviral regimen containing tenofovir disoproxil fumarate plus lamivudine or emtricitabine plus ritonavir-boosted protease inhibitor to a simplified regimen of ritonavir-boosted atazanavir (300/100 mg) plus lamivudine (300 mg) once daily for 48 weeks.
Period: Overall Study
Arm/Group | RTV-Boosted-ATV + 3TC
Started | 31
Completed | 27
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Of the 31 participants enrolled, 1 did not initiate treatment after screening and was excluded from all analyses. Therefore, the baseline and analysis population included 30 participants.
Arm/Group | RTV-Boosted-ATV + 3TC
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [33 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 30
Bone Mineral Density (BMD) at Baseline by DXA [Median (Inter-Quartile Range); unit: g/cm²]
  Lumbar Spine | 0.88 [0.80 to 0.90]
  Left Hip | 0.72 [0.68 to 0.76]

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) at Lumbar Spine and Left Hip From Baseline to Week 48
Description: Mean change in BMD (g/cm²) at lumbar spine (L1-L4) and left hip measured by dual-energy X-ray absorptiometry (DXA) in human immunodeficiency virus-infected adults with hip or spine T-score between < -1.0 and >-2.5
Time Frame: Baseline to Week 48
Measure: Mean (Standard Deviation); unit: g/cm²
Arm/Group | RTV-Boosted-ATV + 3TC
Number analyzed (Participants) | 30
g/cm²
  Lumbar Spine | 0.010 (0.030)
  Left Hip | 0.013 (0.030)
Statistical Analysis 1: Comparison: RTV-Boosted-ATV + 3TC; Single-arm study; no comparator group; Test type: Superiority — Single-arm pilot study to assess BMD improvement after switching therapy. Null hypothesis: no change in lumbar spine BMD at Week 48. Sample size of 45 planned to detect a 2% increase with 90% power (α=0.025). Final analysis included 30 participants; p = 0.0239, Regression, Linear — Statistical test applied to lumbar spine BMD only. P-value reflects within-group change from baseline to Week 48; Per-protocol analysis; missing data excluded; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [0.001 to 0.019], Standard Deviation 0.03 — Represents mean change in lumbar spine BMD from baseline to Week 48
Statistical Analysis 2: Comparison: RTV-Boosted-ATV + 3TC; Single-arm study; no comparator group; Test type: Superiority — Single-arm pilot study to assess BMD improvement after switching therapy. Null hypothesis: no change in left hip BMD at Week 48. Sample size of 45 planned to detect a 2% increase with 90% power (α=0.025). Final analysis included 30 participants; p = 0.0046, Regression, Linear — Left hip; Statistical test applied to left hip BMD only. P-value reflects within-group change from baseline to Week 48; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [0.004 to 0.023], Standard Deviation 0.03 — Represents mean change in left hip BMD from baseline to Week 48

2. Secondary Outcome: Proportion of Patients Free of Virologic Failure (Confirmed Viral Load≥ 50 Copies/mL)
Time Frame: 48 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Patients With Adverse Effects
Time Frame: 48 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Bone Turnover Markers in Blood: Urinary N-terminal Telopeptide of Type-1 Collagen
Time Frame: 48 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Bone Turnover Markers in Blood: Bone-specific Alkaline Phosphatase
Time Frame: 48 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Renald Disfunction Parameter: Estimated Glomerular Filtration Rate
Time Frame: 48 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Renald Disfunction Parameter: Phosphorus in Blood Sample
Time Frame: 48 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: Glucose in Urine
Time Frame: 48 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: Protein in Urine Samples
Time Frame: 48 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: Albumin in Urine Samples
Time Frame: 48 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: Creatinin in Urine Samples
Time Frame: 48 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: Phosphorus in Urine Samples
Time Frame: 48 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: Beta-2 Microglobulin in Urine Samples
Time Frame: 48 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Renald Disfunction, Tubule Dysfunction, Parameter: N-Acetyl-β-D Glucosaminidase in Urine Samples
Time Frame: 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From informed consent to Week 48 (end of study visit)
Description: Adverse events were collected from the time of informed consent until the final study visit (Week 48). Severity was graded using the AIDS Clinical Trial Group (ACTG) Grading Scale. All AEs were recorded regardless of suspected relationship to study drug. Serious adverse events were defined per ICH-GCP guidelines.
Arm/Group | RTV-Boosted-ATV + 3TC
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTV-Boosted-ATV + 3TC (N=30)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This pilot study had a small sample size and did not reach the planned enrollment of 45 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT02652793/Prot_SAP_000.pdf